CLINICAL TRIAL: NCT06940895
Title: Evaluating the Safety and Efficacy of Topical Sirolimus 0.2% to Treat Acanthosis Nigricans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Narrows Institute for Biomedical Research (Other)
Collaborators: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1814310
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-04

CONDITIONS: Acanthosis Nigricans
Keywords: acanthosis nigricans
MeSH Terms: conditions — Acanthosis Nigricans

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patients with Acanthosis Nigricans (Experimental): Patients with the diagnosis of acanthosis nigricans
  Interventions: Drug: Sirolimus 0.2%

INTERVENTIONS:
Drug: Sirolimus 0.2% — sirolimus 0.2% gel
  Other Names: HYFTOR

SUMMARY:
The purpose of this study is to demonstrate the safety and efficacy of Sirolimus 0.2% topical gel for patients with Acanthosis Nigricans

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18+.
* Clinical diagnosis of acanthosis nigricans.
* Available and willing to comply with study instructions and attend all study visits.
* Able and willing to provide written and verbal informed consent.

Exclusion Criteria:

* Subject has any skin pathology or condition that could interfere with the evaluation of the test products or requires the use of interfering topical or systemic therapy.
* Subject has any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in this research study.
* Pregnant, lactating, or is planning to become pregnant during the study.
* Subject is currently enrolled in an investigational drug or device study.
* Subject has received an investigational drug or has been treated with an investigational device within 30 days prior to the initiation of treatment (baseline).
* Subject is unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function.
* Subject has known hypersensitivity or previous allergic reaction to any of the active or inactive components of the test articles.
* Subject has the need or plans to be exposed to artificial tanning devices or excessive sunlight during the trial.
* Erosions, ulcers, or other skin lesions within or closely neighboring the AN lesion application site.
* Hypersensitivity reactions such as anaphylaxis or angioedema to sirolimus or any component of sirolimus 0.2% topical gel (HYFTOR).
* Dyslipidemia (cholesterol level >300mg/dL or >7.75mmol/L, triglyceride level >300 mg/dL or >3.42 mmol/L).
* Subject cannot agree to take appropriate contraception for the duration of the study and 12 weeks after the final dose.
* Exclusions apply to those who have used the following topical treatments to treat AN: retinoids, hydroquinones, corticosteroids, or other depigmenting agents within one month prior to the study, or oral retinoids within six months prior to the study, or medications with mammalian target of rapamycin(mTOR) inhibitory action within 12 months prior to the first visit.
* Subjects with a malignant tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Improvement in hyperpigmentation in acanthosis nigricans lesions | From enrollment to end of treatment at 12 weeks
  Improvement in the Melanin(M) index from baseline to 12 weeks of treatment. The M index is positively correlated with a darker skin color and ranges from 0-999.

SECONDARY OUTCOMES:
Improvement in hyperpigmentation and skin texture in acanthosis nigricans lesions | Baseline to weeks 4, 8, and 12
  Improvement in the ANSC (Acanthosis Nigricans Scoring Chart) from baseline (Day 0) to Visit 2 (Week 4), Visit 3 (Week 8) and Visit 4 (Week 12). ANSC is scored on a scale of 1 to 8 for skin color and 1 to 6 for skin texture. These scores are then combined for a total ANSC score ranging from 2 to 14.
Improvement in the Investigators Global Evaluation (IGE) scale and Patient Global Evaluation (PGE) scale | Baseline to weeks 4, 8, and 12
  IGE and PGE are both scored on a 0 to 6 scale: 0 signifies "clear," 1 indicates "almost clear or > 90% improvement," 2 represents "marked improvement or 75% improvement," 3 denotes "moderate improvement or 50% improvement," 4 signifies "mild improvement or 25% improvement," 5 indicates "no change," and 6 means "worsening."
Improvement in the Dermatology Quality of Life (DLQI) scale | From enrollment to end of treatment at 12 weeks
  The DLQI ranges from 0 to 30 with higher scores denoting worse quality of life.
Assessment of patient satisfaction using the Treatment Satisfaction Questionnaire for Medication (TSQM) | Week 12
  Assessment of patient satisfaction using the treatment satisfaction questionnaire for medication
Digital photography with a TwinFlash RL Clinical Camera to depict clinical improvement of acanthosis nigricans. | Baseline to weeks 4, 8, and 12
  Digital photography with a TwinFlash RL Clinical Camera to depict clinical improvement of AN

CONTACTS AND LOCATIONS:
Overall Officials: Jared Jagdeo, MD MS, Principal Investigator — SUNY Downstate Health Sciences University Department of Dermatology
Locations (1):
- New York Harbor VA Brooklyn Campus, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
undecided whether IPD will be shared.

REFERENCES:
- [Background] Romo A, Benavides S. Treatment options in insulin resistance obesity-related acanthosis nigricans. Ann Pharmacother. 2008 Jul;42(7):1090-4. doi: 10.1345/aph.1K446. Epub 2008 May 20. PMID 18492785
- [Background] Ding X, Bloch W, Iden S, Ruegg MA, Hall MN, Leptin M, Partridge L, Eming SA. mTORC1 and mTORC2 regulate skin morphogenesis and epidermal barrier formation. Nat Commun. 2016 Oct 27;7:13226. doi: 10.1038/ncomms13226. PMID 27807348
- [Background] Dodds M, Maguiness S. Topical sirolimus therapy for epidermal nevus with features of acanthosis nigricans. Pediatr Dermatol. 2019 Jul;36(4):554-555. doi: 10.1111/pde.13833. Epub 2019 Apr 15. PMID 30983034
- [Background] Treesirichod A, Thaneerat N, Kangvanskol W. A comparison of the efficacy and safety profiles of 10% salicylic acid and 10% urea creams in treating acanthosis nigricans in adolescents: a randomized double-blinded study. Arch Dermatol Res. 2023 Sep;315(7):2091-2097. doi: 10.1007/s00403-023-02605-6. Epub 2023 Mar 21. PMID 36943434
- [Background] Pirgon O, Sandal G, Gokcen C, Bilgin H, Dundar B. Social anxiety, depression and self-esteem in obese adolescent girls with acanthosis nigricans. J Clin Res Pediatr Endocrinol. 2015 Mar;7(1):63-8. doi: 10.4274/jcrpe.1515. PMID 25800478
- [Background] Patel NU, Roach C, Alinia H, Huang WW, Feldman SR. Current treatment options for acanthosis nigricans. Clin Cosmet Investig Dermatol. 2018 Aug 7;11:407-413. doi: 10.2147/CCID.S137527. eCollection 2018. PMID 30122971